CLINICAL TRIAL: NCT02449109
Title: Nano Drug Interventional Therapy Using Digital Subtraction Angiography（DSA） for Liver Carcinoma：Clinical Trial
Brief Title: Nano Drug Interventional Therapy Using Digital Subtraction Angiography（DSA） for Liver Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nano drug liver cancer
Record Dates: First submitted 2015-05-14; First posted 2015-05-20 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2015-06

CONDITIONS: Liver Cancer
Keywords: Liver Cancer; Nano drug
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Liver cancer patients never received any interventional therapy.
- Nano drug (Experimental): Liver cancer patients received nano drug interventional therapy using digital subtraction angiography（DSA）. The nano drug is made by mixing Gemzar® with Compound Glycyrrhizin Injection.
  Interventions: Procedure: interventional therapy
- Drug microspheres (Active Comparator): Liver cancer patients received drug microspheres (HepaSphere Microspheres) interventional therapy using digital subtraction angiography（DSA）.
  Interventions: Procedure: interventional therapy

INTERVENTIONS:
Procedure: interventional therapy — Liver cancer patients received drug interventional therapy using the digital subtraction angiography（DSA）
  Arms: Drug microspheres; Nano drug

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of nano drug（Gemzar® mix with Compound Glycyrrhizin Injection） interventional therapy using digital subtraction angiography（DSA） for liver cancer.

DETAILED DESCRIPTION:
By enrolling patients with liver cancer adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of nano drug interventional therapy using digital subtraction angiography（DSA）for liver cancer.

The nano drug is made by mixing Gemzar® with Compound Glycyrrhizin Injection. The nano drug's size is detected by laser diffraction particle size analyzer.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-80
2. Karnofsky performance status >60
3. Diagnosis of liver cancer based on histology or the current accepted radiological measures.
4. Classification tumor,nodes,metastasis-classification(TNM) stage: Ⅱ,Ⅲ,Ⅳ
5. Will receive interventional therapy
6. Life expectancy: Greater than 3 months
7. Patients' routine blood test, liver function and kidney function have no obvious abnormalities
8. Ability to understand the study protocol and a willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients with other primary tumor except liver cancer
2. History of coagulation disorders or anemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse events | 1 year

SECONDARY OUTCOMES:
Percentage of lesions that show no sign of recurrence 12 months after interventional therapy | 1 year
Progress free disease (PFS) | 1 year
Overall survival (OS) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Niu, PhD, Study Chair — Fuda Cancer Hospital
Locations (1):
- Central laboratory in Fuda cancer hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Niu L, Chen J, Yao F, Zhou L, Zhang C, Wen W, Bi X, Hu Y, Piao X, Jiang F, Zeng J, Liu W, Li J, He L, Mu F, Zuo J, Xu K. Percutaneous cryoablation for stage IV lung cancer: a retrospective analysis. Cryobiology. 2013 Oct;67(2):151-5. doi: 10.1016/j.cryobiol.2013.06.005. Epub 2013 Jun 24. PMID 23806858
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Piao+xianghao